CLINICAL TRIAL: NCT03170765
Title: Comparison of Three Different Schedules of Measles Vaccination in Infants: a Pilot Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of Measles Vaccination Schedule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, MAKAM LAXMI GOPAL, JUNIOR RESIDENT, DEPARTMENT OF PEADIATRICS, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LM/PED/01
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: MEASLES DISEASE
MeSH Terms: conditions — Measles | interventions — Measles Vaccine

STUDY DESIGN:
Intervention Model Description: THREE ARM RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are infants ranging from 6-9 months of age. They are expected to be unaware of the intervention. The laboratory personnel performing the antibody level measurements will be blinded by sending the samples with only a four digit code that does not reveal the intervention received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A (Experimental): measles vaccine at 6 months and 9 months of age
  Interventions: Biological: Measles vaccine
- GROUP B (Experimental): measles vaccine at 7.5 months and 9 months of age
  Interventions: Biological: Measles vaccine
- GROUP C (Active Comparator): measles vaccine at 9 months of age (current practice)
  Interventions: Biological: Measles vaccine

INTERVENTIONS:
Biological: Measles vaccine — Live attenuated measles vaccine of brands currently being used in National Immunization Schedule of India.

SUMMARY:
Measles is a preventable infectious viral disease. Since 1985, India has been administering a single dose of measles vaccine to all infants at 9 months of age. This age was chosen to balance the disappearance of maternal (transplacental) antibodies with the increasing risk of developing measles. Thus infants are expected to get protection against measles by acquired maternal measles antibodies derived trans-placentally from the mother for the first 9 months of life. Thereafter vaccine-induced antibodies are expected to protect infants. Seroconversion after measles vaccination does not take place as long as maternal measles antibodies persist in the infant. However, it is widely recognized that a substantial proportion of measles infection (10 to 15%) can occur among infants before the age of measles vaccination. Further, two small cohort studies done in our institution confirm that the majority of infants lose maternal antibodies by six months of age, making them susceptible to measles.This argues strongly for anticipating measles vaccination to an earlier age. However, such early vaccination has the risk that residual maternal antibodies (even if insufficient to protect infants) can neutralize the antigen in the vaccine, rendering vaccination ineffective. Therefore, a careful balance has to be chosen so that low levels of circulating maternal antibodies do not interfere with infants' response to vaccination. However, there is no prospective study in Indian infants to determine the seroconversion and sero-protection rate of earlier vaccination.

This study has following aims and objectives:

1. To study the level of measles specific immunoglobulin G (IgG) antibodies in a cohort of term infants followed from birth to 9 months of age; and the pattern of antibody decline in them.
2. To compare the levels of antibodies in infants at these time points and correlate the levels with the antibody level in the respective mothers at the time of delivery.
3. To compare the efficacy and safety of three different measles vaccination schedules in a cohort of term infants viz (i) vaccination at 9 months of age (current practice), (ii) vaccination at 7.5 months and 9 months of age, and (iii) vaccination at 6 months and 9 months of age.

DETAILED DESCRIPTION:
Study design:

This study has two design components viz.

* Prospective enrollment of a cohort of term infants at birth; and 3 monthly follow-up at the ages of 3 months, 6 months, 9 months and 12 months.
* Randomization at 6 months of age to three intervention groups viz (i) measles vaccination at 9 months of age (as per current practice), (ii) vaccination at 7.5 months and 9 months of age, and (iii) vaccination at 6 months and 9 months of age.

Methods: Enrollment:

Pregnant women awaiting delivery in the Department of Obstetrics and Gynecology will be screened for eligibility (as per the Inclusion and Exclusion criteria). Women whose infants are likely to be eligible for participation in the study will be explained about the nature and purpose of the study prior to delivery. They will be informed about the study protocol and invited to participate. After delivery, mothers and their respective newborn babies, will be enrolled with written, informed consent.

Procedure:

A brief interview will be conducted to determine history of exanthematous illness suffered in the past by the mother, family history of similar illness and vaccinations received by her.

At delivery, approximately 1 ml of cord blood from the infant's side will be collected in a sterile plastic screw-capped container, labeled and transported to the laboratory. Similarly 1 ml of venous blood will be obtained from the mother in a sterile plastic screw-capped container, labeled and transported to the laboratory. Serum will be separated from these samples by centrifugation and deep frozen at minus 20 degree C until analysis.

The infants will be followed-up and undergo venipuncture under aseptic precautions to withdraw 0.8-1.0 ml blood at five further visits viz. 3 months±2 weeks [corresponding to a visit for 2nd/3rd dose of diphtheria- pertussis- tetanus (DPT) vaccine and live oral poliovirus vaccine(OPV)], 6 months±2 weeks (corresponding to visit for 3rd dose of Hepatitis B at 6 months of age), 7.5 months ±2 weeks, at 9 months ±2 weeks (corresponding to visit for measles vaccine as per the current schedule), and at 12 ± 2 weeks months of age (corresponding to visit for routine follow-up).

During the follow-up visit at 6 months of age, infants will be randomized (as described below) to one of three groups viz: Group A: vaccination at 6 months and 9 months of age; Group B: vaccination at 7.5 months and 9 months of age; and Group C: vaccination at 9 months of age (current practice).

Generation of random sequence: A computer programme will be used to generate a random number sequence to allocate participants into three groups in a ratio of 1:1:1, as per the Groups described above.

Allocation concealment: The allocation of each infant will be placed in sealed, opaque envelopes. For each infant presenting at six months of age, one envelope will be marked with the infant's name and then opened. At this stage, the sealed envelopes will contain one of two options viz (i) Vaccination at 6 months or (ii) No vaccination at 6 months. Those who receive the former will follow the protocol for Group A described below. Those who receive the latter will be followed-up at 7.5 months of age; at which stage a second set of sealed enveloped will be accessed. One envelope will be marked with the infant's name and then opened. At this stage, the sealed envelopes will contain one of two options viz (i) Vaccination at 7.5 months or (ii) Vaccination at 9 months. Those who receive the former will follow the protocol for Group B described below; and those who receive the latter will follow the protocol for Group C described below.

Blinding: In this randomized trial design, no attempt will be made to blind the infants being randomized, or their parents (in order to avoid unnecessary injections through a double dummy design). The investigator involved in randomizing the infants will also not be blinded. However, the laboratory personnel performing the antibody level measurements will be blinded by sending the samples with only a four digit code that does not reveal the intervention received.Samples during any visit will be withdrawn prior to administration of vaccine(s).

Measles vaccine will be administered as per the protocol described above by trained personnel in the Immunization Room of the Advanced Pediatrics Center. A standard dose of the available preparation will be administered in the dosage of 0.5 ml through the subcutaneous route. Standard post-vaccination precaution viz observation of the infant for 30 minutes after vaccination will be done to observe for any adverse event.

Clinical protocol:

At each visit history will be elicited to detect clinical features compatible with measles in the baby or any other member of the family in the household contact. This includes:

Any person in whom a clinician suspects measles infection, or Any person with fever and maculopapular rash (i.e. non-vesicular) and cough, coryza (i.e. runny nose) or conjunctivitis (i.e. red eyes).

In addition, the investigator will make a monthly telephone call to the family of enrolled infants asking for specific history compatible with the World Health Organization (WHO) case definition for measles, in the infant or any household member. In case such history is elicited, the infant and affected individual will be invited for clinical examination and a sample of blood will be obtained. Serum will be separated as described and immunoglobulin M (IgM) anti-measles antibody will be measured using commercially available ELISA kits as described below.

After each vaccination, parents of vaccinated infants will be requested to complete a Diary for three days, containing a daily record of (i) excessive crying, (ii) poor feeding, (iii) fever, (iv) redness at injection site, (v) swelling at injection site (vi) tenderness/apparent pain at injection site, and (vii) any other unusual behavior/appearance in the infant.

Laboratory processing:

Clotted blood samples will be centrifuged at 3000 rpm for 15 minutes to obtain serum which will be frozen at -20 degree Celsius till tested. Serum will be processed in batches of 30-40 and measles specific IgG antibodies will be quantified by micro-ELISA (enzyme linked immunosorbent assay) using commercially available quantitative measles IgG kits of high sensitivity (98-100%) and specificity (100%). IgM antibody assay will be done to confirm the diagnosis of measles only in those infants suspected to have measles; using commercially available quantitative measles IgG kits of high sensitivity (98-100%) and specificity (100%). Sera from subjects, calibrators, positive and negative controls will be diluted in serum diluents and test will be performed as recommended by the manufacturers. The obtained optical density value for each sample will be converted into measles antibody titre in units/ml with help of calibrator values in a standard log graph paper and these units/ml will then be interpreted as International Units/ml taking the recommendation in the kit.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at term (i.e.> 37 completed weeks of gestation) within the hospital will be eligible for inclusion into the study.

Exclusion Criteria:

1. Infants born to mothers known to have known immunodeficiency determined through examination of clinical records (HIV positive and those on immunosuppressive therapy during pregnancy).
2. Babies born with antenatally or postnatally diagnosed congenital anomalies that are anticipated to be life-threatening.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of protected infants from measles. | 6 weeks after vaccination
  Infants with serum anti measles IgG antibody levels higher than 200 m IU/ml, or other specific values provided by manufacturers in the antibody kits, will be taken as protected.

SECONDARY OUTCOMES:
Incidence of treatment - emergent adverse events | 3 days after vaccination
  This will be done by calculation of proportion of infants who develop any of the following features : 1. Excessive crying and poor feeding ; 2. Fever; 3. Redness or swelling at injection site; 4. Tenderness/apparent pain at injection site; 5. Any other unusual behaviour/appearance in infant. The presence of each event on a given day will be given a score of 1. The total score for all three days will be added to get a composite Safety score. In addition, any adverse event (AE) or serious adverse event (SAE) occurring within 30 minutes of vaccination (as per standard protocol) will be recorded.
  Event Day 1 Day 2 Day 3 Excessive crying Poor feeding Fever Redness at injection site Swelling at injection site Tenderness/apparent pain at injection site Any other unusual behavior/appearance in the infant Total score
Infant- Mother antibody correlation at birth | At birth
  Correlation of infant antibody levels at birth with maternal antibody levels
Infant- Mother antibody correlation at 3 months | At 3 months of age
  Correlation of infant antibody levels at 3 months of age with maternal antibody levels
Infant- Mother antibody correlation at 6 months | At 6 months of age
  Correlation of infant antibody levels at 6 months of age with maternal antibody levels
Susceptibility among not vaccinated infants | Birth to 12 months of age
  Proportion of not vaccinated infants susceptible to measles at birth, 3 months, 6 months, and 9 months of age
Susceptibility among vaccinated infants | Birth to 12 months of age
  Proportion of vaccinated infants susceptible to measles at birth, 3 months, 6 months, 9 months, and 12 months of age; and correlation to vaccination status
Acute measles | Birth to 12 months of age
  Proportion of infants who develop acute measles infection and correlation to vaccination status

CONTACTS AND LOCATIONS:
Overall Officials: LAXMI MAKAM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; JOSEPH L MATHEW, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh; SOURABH DUTTA, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; VANITA SURI, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; R K RATHO, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; BHAVNEET BHARTI, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; MINI P SINGH, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared with institutional ethics committee on request.